CLINICAL TRIAL: NCT07186751
Title: Comparing the Efficacy and Safety of Pregabalin Monotherapy With Pregabalin Combined Other Neuromodulatory Drugs (Venlafaxine) in the Treatment of Fibromyalgia: A Multicenter Clinical Study
Brief Title: The Efficacy and Safety of Pregabalin Combined With Venlafaxine in Patients With Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: China-Japan Friendship Hospital (Other); First Affiliated Hospital of Army Medical University, PLA (Unknown); Second Affiliated Hospital of Guangxi Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director, Department of Pain Management, Principal Investigator, Clinical Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-217-03-03
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia; Pregabalin; Venlafaxine; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Pregabalin; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin monotherapy group (Active Comparator)
  Interventions: Drug: Pregabalin
- Pregabalin with venlafaxine group (Experimental)
  Interventions: Drug: Pregabalin with venlafaxine

INTERVENTIONS:
Drug: Pregabalin — In general, for the pregabalin monotherapy group (Pregabalin Capsules, Pfizer, New York, USA), treatment will be initiated at 150 mg/day, administered in two divided doses. After 7 days, the dose will be increased to 300 mg/day. Thereafter, based on individual response and tolerability, the dose may be further increased to a maximum of 450 mg/day.
  Arms: Pregabalin monotherapy group
Drug: Pregabalin with venlafaxine — For the combination therapy group, participants will receive both pregabalin and venlafaxine (Venlafaxine Hydrochloride Sustained-Release Capsules, Pfizer, Co Kildare, Ireland). The dose titration for pregabalin will be identical to that of the monotherapy group. Concurrently, venlafaxine will be initiated at 75 mg/day. If well-tolerated, the dose may be increased in 75 mg/day increments at weekly intervals, guided by clinical response and side effects profile, to a maximum dose of 225 mg/day.
  Arms: Pregabalin with venlafaxine group

SUMMARY:
Fibromyalgia (FM) is a chronic pain syndrome characterized by widespread pain, fatigue, and emotional disorders. Its onset is related to factors such as central sensitization and imbalance of neurotransmitters. The current mainstream treatments include pregabalin, but the efficacy of pregabalin is limited, with only 25%-40% pain relief rate, and adverse reactions are common. Selective serotonin and norepinephrine reuptake inhibitors (SNRIs), such as duloxetine, has demonstrated efficacy in FM by modulating pain pathways through increased serotonin and norepinephrine availability. Several studies have highlighted benefits of venlafaxine in FM. We hypothesize that the combination of pregabalin with venlafaxine may offer greater pain relief compared pregabalin monotherapy, without a significant increase in adverse effects for patients with FM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with FM according to the 2016 Revisions to the 2010/2011 FM diagnostic criteria;
* Aged more than 18 years;
* Suffering from moderate to severe FM with 11-point numeric rating scale (NRS) score more than 4 at baseline that have not been effectively alleviated by non-pharmacological treatments and has not received currently recommended pharmacological treatment for FM;
* Agreed to sign the informed consent form.

Exclusion criteria

* A history of psychiatric disease;
* Hypersensitivity or have contraindications to pregabalin, venlafaxine;
* Pregnancy or breastfeeding;
* Presence of serious systemic diseases, including uncontrolled hypertension, uncontrolled diabetes, significant cardiac dysfunction, or chronic hepatic or renal dysfunction;
* With acute or chronic pain conditions other than FM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
The average pain intensity | At the 4-weeks
  The average pain intensity over the past 24 hours, rated each morning upon awakening and averaged over 7 days at the 4 weeks. This will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.

SECONDARY OUTCOMES:
The worst pain intensity | At the weeks 1, 2, 4, 8, and 12
  The worst pain intensity over the past 24 hours, rated each morning upon awakening and averaged over 7 days. The pain intensity will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.
The proportion of patients achieving pain reduction | At the weeks 1, 2, 4, 8, and 12
  The proportion of patients achieving a ≥ 50% and ≥ 30% reduction in mean baseline pain intensity. The pain intensity will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.
Dose of pregabalin and/or venlafaxine | At the weeks 1, 2, 4, 8, and 12
  At the aforementioned follow-up time points, the researchers will inquire about the current dosages of pregabalin and/or venlafaxine being administered to the participants. Any dose adjustments, interruptions, or discontinuations, along with the reasons will be documented in detail.
The Revised FM Impact Questionnaire | At the weeks 1, 2, 4, 8, and 12
  The Revised FM Impact Questionnaire assesses the severity of FM symptoms and their impact on daily functioning. It evaluates three linked domains: function, overall impact, and symptoms, using a 0 to10 NRS. The total score ranges from 0 to 100, with higher scores indicating greater disease burden.
The Brief Pain Inventory (BPI) severity (BPI-S) and interfere (BPI-I) subscales | At the weeks 1, 2, 4, 8, and 12
  BPI-S accesses pain intensity over the past 24 hours, calculated as the average of items 3 to 6 on the BPI, scored using a 0 to 10 NRS. In the NRS scale, 0 indicates no pain, while 10 represents the worst pain imaginable. The total score ranges from 0 to 40, with higher scores indicating greater pain severity. BPI-I evaluates the degree to which pain interferes with daily activities, including general activity, mood, mobility work, relationships, sleep, and pleasure. This subscale comprises 7 items, each scored from 0 (no interference) to 10 (complete interference), with a total score ranging from 0 to 70.
The short-form 36 Health Survey (SF-36) | At the weeks 1, 2, 4, 8, and 12
  The SF-36 assesses health-related quality of life, capturing preferences across various health states. It assesses 8 dimensions: physical functioning, physical role limitations due to physical health, bodily pain, general health, vitality, social functioning, emotional role limitations due to emotional problems, and mental health. Scores range from 0 to 100 for each dimension, with higher scores indicating better health status.
The Medical Outcomes Study Sleep Scale (MOS) | At the weeks 1, 2, 4, 8, and 12
  The MOS is a questionnaire comprising 12 items that assess various aspects of sleep using a 6-point ordinal scale (1 indicating permanence and 6 indicating absence).
The Beck Depression Inventory-Ⅱ (BD-Ⅱ) | At the weeks 1, 2, 4, 8, and 12
  The BD-Ⅱ evaluates the severity of depressive symptoms using a 4-point scale from 0 to 3, where 0 indicates no symptom and 3 indicates severe symptomatology. It comprises 21 items, the total score ranging from 0 to 63.
Adverse Events | Through study completion, an average of 12 weeks
  The incidence and proportion of adverse events will be recorded and categorized as mild, moderate, severe, or life-threatening. AEs are defined as events that arise during treatment, were absent before treatment, or worsen relative to the pretreatment state.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Beijing, Beijing 100070, Beijin
  - Beijing Tiantan Hospital, Beijing, Beijing 100070, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) are available. Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.

REFERENCES:
- See also: Mathieson S, Lin C-WC, Underwood M, Eldabe S. Pregabalin and gabapentin for pain. BMJ. 2020;369:m1315. doi: 10.1136/bmj.m1315 — https://pubmed.ncbi.nlm.nih.gov/32345589/
- See also: Migliorini F, Maffulli N, Eschweiler J, Baroncini A, Bell A, Colarossi G. Duloxetine for fibromyalgia syndrome: a systematic review and meta-analysis. J Orthop Surg Res. 2023;18(1):504. doi: 10.1186/s13018-023-03995-z. — https://pubmed.ncbi.nlm.nih.gov/37461044/
- See also: Gilron I, Chaparro LE, Tu D, Holden RR, Milev R, Towheed T, et al. Combination of pregabalin with duloxetine for fibromyalgia: a randomized controlled trial. Pain. 2016;157(7):1532-40. doi: 10.1097/j.pain.0000000000000558. — https://pubmed.ncbi.nlm.nih.gov/26982602/
- See also: VanderWeide LA, Smith SM, Trinkley KE. A systematic review of the efficacy of venlafaxine for the treatment of fibromyalgia. J Clin Pharm Ther. 2015;40(1):1-6. doi: 10.1111/jcpt.12216. — https://pubmed.ncbi.nlm.nih.gov/25294655/